CLINICAL TRIAL: NCT00755794
Title: An 8 Week Multicenter, Open-label, Observational Study to Evaluate the Effectiveness of Adding Montelukast Sodium 10 mg Per Day to Inhaled Corticosteroids in Adult Subjects With Uncontrolled Asthma
Brief Title: The Singulair® add-on Study Effectiveness of Adding Montelukast to Inhaled Corticosteroids in Adult Subjects With Uncontrolled Asthma (0476-384)
Acronym: SAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0476-384; 2008_548
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2024-06-07 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

ARMS (1):
- 1 (Experimental): Montelukast
  Interventions: Drug: montelukast sodium

INTERVENTIONS:
Drug: montelukast sodium — Montelukast Tablet, 10 mg, 8 weeks, daily
  Other Names: Singulair

SUMMARY:
The purpose of this study is to evaluate the effectiveness of adding Montelukast Sodium (singulair®) 10 mg per day to inhaled corticosteroids in adult subjects with uncontrolled asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients Is 18 Years Old

Note 1: Regulatory Requirements Necessitate The Following Criterion. It May Not Be Appropriate For Your Patients. Female Patients Of Childbearing Potential Should Be Informed Not To Become Pregnant During The Study By Using The Appropriate Contraceptive Methods (Oral Or Long-Acting Contraceptive Injections (Depo Provera), Intrauterine Device (Iud), Or Barrier Methods (E.G. Condom Or Diaphragm Plus Spermicide) Or To Be Abstinent (No Sexual Intercourse)) Beginning At Least 7 Days Before Visit 1 And Continuing At Least 14 Days After Visit 4 Or A Discontinuation Visit

Note 2: For Alberta: Investigators Who Will Recruit In Private Office, No Patients Can Be Recruited In The Study Until Approval From The College Of Physicians And Surgeons Of Alberta Ethics Committee Is Obtained

Exclusion Criteria:

* Patient Is Well Controlled, Adherent And Satisfied With Current Controller Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2006-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To describe the percentage of patients with asthma who will be controlled after 8 weeks of treatment with montelukast used in combination with inhaled corticosteroids | 8 weeks

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of montelukast | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] FitzGerald JM, Foucart S, Coyle S, Sampalis J, Haine D, Psaradellis E, McIvor RA. Montelukast as add-on therapy to inhaled corticosteroids in the management of asthma (the SAS trial). Can Respir J. 2009 May-Jun;16 Suppl A(Suppl A):5A-14A. doi: 10.1155/2009/593753. PMID 19557206
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html